CLINICAL TRIAL: NCT06432348
Title: Pilates Exercises and Soccer: A Comparative Study of Mat vs. Reformer on FMS and ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Osman Yılmaz, PhD, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OsmaniyeKAU Osman Yılmaz
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sports, Mechanical
Keywords: Functional movement screening; Mat pilates; Reformer pilates; Range of motion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reformer Pilates (Experimental): Before starting the exercises, a 5-minute warm-up session was performed. The reformer Pilates exercise program included movements such as the Footwork Series (Toes, Heels, Tendon Stretch, V Position), Supine Arm Series (Pull, Circle, Pull Head Up, Triceps Press), Short Box Series (Round, Flat Back, Twist), Short Box and Arm Series (Chest Fly, The Gift, Rhomboid, Biceps Curl, Rowing, Triceps), Long Box Series (Swan, Pulling Fly), Stomach Massage (Round, Twist), Knee Stretch (Round, Flat Back), Hip Work Series (Double Leg Press, Hamstring Pulls, Leg Circle, Frog), Elephant, and Side Stretch. Participants had two-minute rest intervals after the Supine Arm Series, Short Box, Arm Series, and Knee Stretch movements. Movements were performed with ten repetitions in the first four weeks and 12 repetitions in the following four weeks.
  Interventions: Other: Reformer pilates
- Mat Pilates (Experimental): Before the exercises, a 5-minute warm-up session was performed. The mat Pilates exercise program included movements such as Rol Up, One Leg Circle, Double Leg Straight Lower, One Leg Stretch, Criss Cross, Toe Top, Shoulder Bridge, Seated Tracking, Spine Twist, Up-Down Side Kick, Front-Back Side Kick, Circle Side Kick, Flight, Swan, Rest Position, Swimming, Push Up, Long Stretch, Cat Cow, Mermaid Stretch. The participants had two-minute rest breaks after the toe-top, spine twist, and circle side-kick movements. Movements were performed with ten repetitions in the first four weeks and 12 repetitions in the following four weeks.
  Interventions: Other: Mat Pilates
- Control (No Intervention)

INTERVENTIONS:
Other: Reformer pilates — Before starting the exercises, a 5-minute warm-up session was performed. The reformer Pilates exercise program included movements such as the Footwork Series (Toes, Heels, Tendon Stretch, V Position), Supine Arm Series (Pull, Circle, Pull Head Up, Triceps Press), Short Box Series (Round, Flat Back, Twist), Short Box and Arm Series (Chest Fly, The Gift, Rhomboid, Biceps Curl, Rowing, Triceps), Long Box Series (Swan, Pulling Fly), Stomach Massage (Round, Twist), Knee Stretch (Round, Flat Back), Hip Work Series (Double Leg Press, Hamstring Pulls, Leg Circle, Frog), Elephant, and Side Stretch. Participants had two-minute rest intervals after the Supine Arm Series, Short Box, Arm Series, and Knee Stretch movements. Movements were performed with ten repetitions in the first four weeks and 12 repetitions in the following four weeks. The participants underwent six weekly training sessions over eight weeks, comprising three Reformer Pilates sessions and three team training days.
  Arms: Reformer Pilates
Other: Mat Pilates — Before the exercises, a 5-minute warm-up session was performed. The mat Pilates exercise program included movements such as Rol Up, One Leg Circle, Double Leg Straight Lower, One Leg Stretch, Criss Cross, Toe Top, Shoulder Bridge, Seated Tracking, Spine Twist, Up-Down Side Kick, Front-Back Side Kick, Circle Side Kick, Flight, Swan, Rest Position, Swimming, Push Up, Long Stretch, Cat Cow, Mermaid Stretch. The participants had two-minute rest breaks after the toe-top, spine twist, and circle side-kick movements. Movements were performed with ten repetitions in the first four weeks and 12 repetitions in the following four weeks. Movements were performed with ten repetitions in the first four weeks and 12 repetitions in the following four weeks. The participants underwent six weekly training sessions over eight weeks, comprising three Mat Pilates sessions and three team training days.
  Arms: Mat Pilates

SUMMARY:
Pilates exercises have been used to improve core strength, trunk and shoulder strength, lower body strength, agility, dynamic balance, coordination skills, flexibility, and posture in various sports. A previous study demonstrated the beneficial impact of mat Pilates exercises on the functional performance of soccer players. However, more research is needed to understand the effects of Pilates on the FMS and ROM. Consequently, this study aimed to investigate and compare the influence of mat Pilates and reformer Pilates exercises on FMS and ROM in soccer players, addressing this critical research gap.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults 19 to 20 years old
* Gender: Male
* Volunteering players

Exclusion Criteria:

- Diagnosis: Diagnosis of a specific medical condition

Ages: 19 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screening and range of motion tests | One week
  Thirty voluntary participants were randomly assigned to either RP (n=10; mean age = 20.60 ± 1.65), MP (n=10; mean age = 19.40 ± 1.35), or CG (n=10; mean age = 20.10 ± 1.15). The Functional Movement Screening Test Kit was used in this study. It consists of seven movements: Deep Squat, Hurdle Step, In-Line Lunge, Shoulder Mobility, Active Straight Leg Raise, Trunk Stability Push-Up, and Rotary Stability. Each test was scored on a scale ranging from 0 to 3, with the highest possible score being 21 . Based on previous research, participants with a total FMS score lower than 14 were considered to have a higher risk of injury.
Range of motion tests | One week
  Thirty voluntary participants were randomly assigned to either RP (n=10; mean age = 20.60 ± 1.65), MP (n=10; mean age = 19.40 ± 1.35), or CG (n=10; mean age = 20.10 ± 1.15). Joint range of motion measurements were made to evaluate the joint range of motion of the athletes. Tests were conducted: shoulder hyperextension, hip flexion, hip extension, hip abduction, hip internal rotation, hip external rotation, ankle dorsiflexion, and ankle plantar flexion. Joint range of motion measurement was performed with a goniometer.Measurements were recorded in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No